CLINICAL TRIAL: NCT06499220
Title: Electrically Evoked Compound Action Potentials Human Observation Medtronic System Study (ECHO-MDT)
Acronym: ECHO-MDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT19014
Record Dates: First submitted 2024-06-18; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ECAP Recording (Experimental)
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — Spinal Cord Stimulation (SCS) as an aid in the management of chronic, intractable pain of the trunk and/or limbs.

SUMMARY:
This is a prospective, multi-center, non-significant risk IDE study of evoked waveforms resulting from stimulation of the dorsal column using a closed-loop system. comprised of Medtronic hardware or off the shelf hardware, which uses recorded waveforms to adjust stimulation amplitude.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older
2. Candidate for or undergoing Medtronic SCS device trial for labeled indication*
3. Willing and able to provide signed and dated informed consent
4. Capable of comprehending and consenting in English
5. Willing and able to comply with all study procedures and visits *Candidate for or undergoing Medtronic SCS device trial for labeled indication means that a clinical decision has already been made between a physician and the patient to undergo Medtronic SCS trialing to treat the patient's chronic pain. This decision is to be made prior to discussing with the patient whether to enroll in the study.

Exclusion Criteria:

1. Implanted electrical cardiac device (e.g., pacemaker, defibrillator)
2. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the Medtronic study manager or designee)
3. Currently diagnosed with a disease that may confound ability to evoke compound action potentials, e.g. multiple sclerosis, as determined by the investigator
4. Pregnant or is of child-bearing potential and unwilling to use a medically acceptable form of birth control during the study
5. Has untreated major psychiatric comorbidity, as determined by the investigator or designee
6. Trialed with a permanent implant lead and extension ("buried lead trial")

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Collection of ECAP data (sensing configurations, stimulation parameters eliciting ECAPs, control policies/algorithms for recording ECAPs) via the research system. | 1 hour to 72 hours
  The ECAP data collected is prototype system/device information for development of a closed loop system.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - MercyOne Des Moines Medical Center, Des Moines, Iowa
  - Nura Research Institute, Edina, Minnesota
  - Twin Cities Pain Clinic, Edina, Minnesota
  - iSpine Pain Physicians, Maple Grove, Minnesota
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Kettering Health, Kettering, Ohio
  - Premier Pain Treatment Institute, Mount Orab, Ohio
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - Rockefeller Neuroscience Institute West Virginia University, Morgantown, West Virginia